CLINICAL TRIAL: NCT01250054
Title: Comparison of Two Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-319-C-018
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2011-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lotrafilcon B / Comfilcon A (Other): Lotrafilcon B multifocal contact lenses worn first, with comfilcon A multifocal contact lenses worn second. Each product worn bilaterally on a daily wear basis for one week.
  Interventions: Device: Lotrafilcon B contact lens; Device: Comfilcon A contact lens
- Comfilcon A /Lotrafilcon B (Other): Comfilcon A multifocal contact lenses worn first, with lotrafilcon B multifocal contact lenses worn second. Each product worn bilaterally on a daily wear basis for one week.
  Interventions: Device: Lotrafilcon B contact lens; Device: Comfilcon A contact lens

INTERVENTIONS:
Device: Lotrafilcon B contact lens — Commercially marketed, silicone hydrogel, multifocal contact lens for daily wear use
  Other Names: AIR OPTIX AQUA MULTIFOCAL
Device: Comfilcon A contact lens — Commercially marketed (Europe), silicone hydrogel, multifocal contact lens for daily wear use
  Other Names: BIOFINITY MULTIFOCAL

SUMMARY:
The purpose of this study is to compare two multifocal contact lenses in presbyopic wearers.

ELIGIBILITY:
Inclusion Criteria:

* At least 35 years of age.
* Sign written Informed Consent
* Spectacle add of +0.50 to +2.50D.
* Best corrected visual acuity of at least 20.30 in both eyes.
* Currently wearing soft contact lenses at least 5 days per week.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks of enrollment.
* Currently enrolled in any clinical trial.
* Astigmatism > 1.00D.
* Strabismus/amblyopia.
* Other protocol-defined exclusion criteria may apply.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This reporting group includes all enrolled and dispensed participants.
Period: Period 1, One Week of Wear
Arm/Group | Lotrafilcon B / Comfilcon A | Comfilcon A /Lotrafilcon B
Started | 8 | 8 (One subject did not wear Period 1 lenses due to power availability and proceeded to Period 2 lenses.)
Completed | 8 (One subject discontinued between Period 1 and Period 2 due to power availability.) | 8 (One subject discontinued between Period 1 and Period 2 due to noncompliance.)
Not Completed | 0 | 0
Period: Period 2, One Week of Wear
Arm/Group | Lotrafilcon B / Comfilcon A | Comfilcon A /Lotrafilcon B
Started | 7 | 8
Completed | 6 | 8
Not Completed | 1 | 0
Not completed — Unacceptable subjective vision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed subjects.
Arm/Group | Overall
Number analyzed (Participants) | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 48.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Vision
Description: Overall vision, as interpreted by the participant and recorded by the investigator as a single, retrospective evaluation of one week's wear time. Overall vision was measured on a 10-point scale, with 1 being worst and 10 being best.
Time Frame: One week of wear
Population: Analysis conducted per protocol, with exclusions due to reasons such as: major protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lotrafilcon B: Commercially marketed, silicone hydrogel, multifocal contact lenses for daily wear use worn bilaterally for one week.
- Comfilcon A: Commercially marketed (Europe), silicone hydrogel, multifocal contact lenses for daily wear use worn bilaterally for one week.
Arm/Group | Lotrafilcon B | Comfilcon A
Number analyzed (Participants) | 16 | 13
units on a scale | 8.5 (1.2) | 8.3 (1.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 19 days.
Description: This reporting group includes all enrolled and exposed participants.
Arm/Group | Lotrafilcon B | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes